CLINICAL TRIAL: NCT03128580
Title: Embryo Aneuploidies and Morphokinetics in Ovarian Stimulated and Non Stimulated Cycles. An Intrapatient Comparison Using Next Generation Sequencing in Biopsy of Blastocysts and Time Lapse Evaluation.
Brief Title: Embryo Aneuploidies and Morphokinetics in Ovarian Stimulated and Non Stimulated IVF Cycles
Acronym: AMOS
Status: Terminated | Type: Observational
Why Stopped: After an interim analysis, it was decided to discontinue the study after a stochastic curtailment analysis.
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1703-VLC-021-EL
Record Dates: First submitted 2017-04-10; First posted 2017-04-25 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Euploid Embryos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural Cycle: The patient will not undergo hyperstimulation rather a natural cycle
- Stimulated Cycle: The 80 patients will undergo hyperstimulation cycle as per the clinical practice planned for the patient.

SUMMARY:
The purpose of this study is to compare the number of euploid embryos obtained per metaphase II oocyte in unstimulated (modified natural cycles) and stimulated IVF cycles.

DETAILED DESCRIPTION:
Effects of ovarian stimulation on human embryo quality is still a subject of study. When natural and stimulated cycles have been compared, no differences have been observed in terms of embryo cleavage capacity, oocyte and embryo aneuploidy rate or incidence of aneuploidy in aborted foetuses. When mild and conventional doses of gonadotropins have been compared, a higher proportion of good morphological quality embryos are observed in the former. On the contrary, we showed that ovarian stimulation does not increase significantly the embryo aneuploidy rate in IVF derived human embryos when unstimulated and stimulated cycles were compared in oocyte donors. In this study, we want to compare the embryo aneuploidy rate between unstimulated and stimulated cycles in infertile patients, subjected to both IVF cycles with blastocyst biopsy and NGS-PGS. A comparison of the morphokinetics will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 30-38 years old (inclusive)
* with regular menstrual cycles (25-35 days)
* AntiMülleriana Hormone >5 pmol/L.
* Undergoing IVF treatment

Exclusion Criteria:

* BMI >30 kg/m2
* repeated miscarriages
* implantation failure
* uterine or adnexal pathology
* Unable to be treated with gonadotrophins for the ovarian hyperstimulation
* history of low response to ovarian hyperstimulation
* participation in another study with PGS for monogenic pathology
* Cryptozoospermia in male partner

Ages: 30 Years to 38 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Women undergoing fertility treatment
Study Population: Women undergoing In Vitro Fertilization treatment
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Comparison of the number of euploid embryos from Metaphase II oocytes in different cohorts of embryos. | 30 days
  Number of metaphase II oocyte per euploid embryo in unstimulated and stimulated cycles.

SECONDARY OUTCOMES:
Incidence of embryo aneuploidies in two cohorts of embryos. | 30 days
  Incidence of embryo aneuploidies between the unstimulated and stimulated cycle in the same patient
Morphokinetic evaluation of embryos in two different cohorts of embryos. | 30 days
  Morphokinetic evaluation of the embryos obtained in an unstimulated and stimulated cycle

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - IVI Valencia, Valencia
  - Instituto Valenciano de Infertilidad Spain, Valencia

IPD SHARING:
Plan to Share IPD: No